CLINICAL TRIAL: NCT04458051
Title: A Phase 3, Randomized, Double-blind, Efficacy and Safety Study Comparing SAR442168 to Placebo in Participants With Primary Progressive Multiple Sclerosis (PERSEUS)
Brief Title: Primary Progressive Multiple Sclerosis (PPMS) Study of Bruton's Tyrosine Kinase (BTK) Inhibitor Tolebrutinib (SAR442168) (PERSEUS)
Acronym: PERSEUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC16035; U1111-1238-1318 (Registry Identifier: ICTRP); 2024-514495-41 (Registry Identifier: CTIS); 2020-000645-14 (EudraCT Number)
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Primary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SAR442168 (Experimental): Dose 1 of oral SAR442168 once daily
  Interventions: Drug: Tolebrutinib
- Placebo (Placebo Comparator): Placebo to match the SAR442168 once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tolebrutinib — Pharmaceutical form: Film-coated Tablet Route of administration: Oral
  Other Names: SAR442168
  Arms: SAR442168
Drug: Placebo — Pharmaceutical form: Film-coated Tablet Route of administration: Oral
  Arms: Placebo

SUMMARY:
Primary Objective:

To determine the efficacy of SAR442168 compared to placebo in delaying disability progression in primary progressive multiple sclerosis (PPMS)

Secondary Objectives:

To evaluate efficacy of SAR442168 compared to placebo on clinical endpoints, magnetic resonance imaging (MRI) lesions, cognitive performance, physical function, and quality of life To evaluate safety and tolerability of SAR442168 To evaluate population pharmacokinetics (PK) of SAR442168 in PPMS and its relationship to efficacy and safety To evaluate pharmacodynamics of SAR442168

DETAILED DESCRIPTION:
Study duration will vary per participant in this event driven trial with a treatment duration of approximately 12 to 60 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 55 years of age inclusive
* Diagnosis of PPMS according to the 2017 McDonald criteria
* Expanded disability status scale (EDSS) score between 2.0 to 6.5 points, at screening inclusive
* Positive cerebrospinal fluid oligoclonal bands and/or elevated Immunoglobulin G (IgG) index either during screening or documented previous history.
* Contraceptive use consistent with local regulations for individuals participating in clinical studies
* Participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:
* Is not a woman of childbearing potential (WOCBP) or is a WOCBP and agrees to use an acceptable contraceptive method
* the participant must not have access to ocrelizumab (eg, ocrelizumab not available on the national market or not reimbursed for the approved indication).
* the participant must have access to and be eligible to be treated with ocrelizumab but: 1) does not tolerate it due to side effects or safety reasons; and/or 2) has failed ocrelizumab treatment due to perceived lack of efficacy

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Participant has conditions that would adversely affect study participation such as short life expectancy.
* Evidence of infection with human immunodeficiency virus (HIV), transplantation, progressive multifocal leukoencephalopathy (PML), active hepatitis B or C, active or latent tuberculosis or other active infection that would adversely affect study participation.
* Persistent chronic or active or recurring system infection that may adversely affect participation or IMP administration in this study as judged by the investigator
* History of malignancy within 5 years prior to screening.
* History of alcohol or drug abuse within 1 year prior to Screening.
* Hospitalized for psychiatric disease within 2 years prior to Screening.
* Clinically significant laboratory abnormalities (including evidence of liver injury) or electrocardiogram abnormalities at Screening.
* A bleeding disorder or known platelet dysfunction at any time prior to the screening visit.
* A platelet count <150 000/μL at the screening visit.
* A history of significant bleeding event within 6 months prior to screening, according to the Investigator's judgment such as, but not limited to cerebral or gastrointestinal
* Lymphocyte count below the lower limit of normal at Screening.
* Recent live (attenuated) vaccine within 2 months before the first treatment visit.
* Recent major surgery (within 4 weeks of Screening) or planned major surgery during the study.
* The participant has received medications/treatments for MS within a specified time frame.
* Receiving potent and moderate inducers of cytochrome P450 3A (CYP3A) or potent inhibitors of CYP2C8 hepatic enzymes.
* Receiving anticoagulant or antiplatelet therapy (such as aspirin >81mg/day, clopidogrel, warfarin).
* Contraindications to magnetic resonance imaging (MRI).

NOTE: Other Inclusion/Exclusion criteria may apply. The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 767 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
6-month composite Confirmed Disability Progression (cCDP) | Up to approximately 60 months
  Time to onset of 6-month cCDP defined as follows:
  Increase over at least 6 months of ≥1.0 point from the baseline expanded disability status scale (EDSS) score when the baseline score is ≤5.5, or ≥0.5 points when the baseline EDSS score is >5.5, or ≥20% from the baseline T25-FW, or ≥20% from the baseline 9-HPT

SECONDARY OUTCOMES:
6-month Confirmed Disability Progression (CDP) | Up to approximately 60 months
  Time to onset of 6-month CDP as assessed by EDSS score
3-month composite Confirmed Disability Progression (cCDP) | Up to approximately 60 months
  Time to onset of 3-month cCDP
Change in T2 hyperintense lesions by MRI | From screening MRI to approximately 60 months
  Total number of new and/or enlarging T2 hyperintense lesions as detected by MRI after baseline up to and including the end of study (EOS)
Time to onset of confirmed disability improvement (CDI) | Up to approximately 60 months
  Time to onset of CDI defined as ≥1.0-point decrease on the EDSS score from baseline confirmed over at least 6 months
Percent change in Brain volume (BV) | From 6 months up to approximately 60 months
  Percent change in brain volume (BV) as detected by brain MRI at the EOS compared to month 6
Change in cognitive function as assessed by SDMT | From Baseline up to approximately 60 months
  Change in cognitive function at the EOS compared to baseline as assessed by the Symbol Digit Modalities Test (SDMT)
Change in cognitive function as assessed by CVLT-II | From Baseline up to approximately 60 months
  Change in cognitive function at the EOS compared to baseline as assessed by the California Verbal Learning Test II (CVLT-II) where available
Change in Multiple Sclerosis Quality of Life | From Baseline up to approximately 60 months
  Change in Multiple Sclerosis Quality of Life-54 (MSQoL-54) at the EOS compared to baseline
Safety and Tolerability | From screening up to approximately 60 months
  Number of participants with adverse events (AEs), Serious AEs, AEs leading to permanent study intervention discontinuation, and adverse events of special interest (AESI)
Population pharmacokinetics | Months 6, 9 and 12
  Plasma concentration of SAR442168 (population PK assessment) at Months 6, 9, and 12
Change in plasma neurofilament light chain (NfL) | From Baseline up to approximately 60 months
  Change in NfL levels from at the EOS compared to baseline
Change in lymphocyte phenotype subsets | From Baseline up to approximately 60 months
  Change in lymphocyte phenotype subsets in whole blood at the EOS compared to baseline in a subset of participants
Changes in serum Immunoglobulin level | From Baseline up to approximately 60 months
  Changes in serum Immunoglobulin level at the EOS compared to baseline
Change in serum chitinase-3 like protein 1 (Chi3L1) | From Baseline up to approximately 60 months
  Change in serum Chi3L1 at EOS compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (277):
- United States (45):
  - UC San Diego ACTRI Site Number : 8400101, La Jolla, California
  - Collaborative Neuroscience Research Site Number : 8400045, Los Alamitos, California
  - Multiple Sclerosis Center- Site Number : 8400143, Los Angeles, California
  - Multiple Sclerosis Center of California Site Number : 8400135, Newport Beach, California
  - SC3 Research - Pasadena Site Number : 8400070, Pasadena, California
  - University of San Francisco, Sandler Neurosciences Center- Site Number : 8400137, San Francisco, California
  - Harbor UCLA Site Number : 8400088, Torrance, California
  - Regina Berkovich, MD, PhD Site Number : 8400059, West Hollywood, California
  - Advanced Neurosciences Research Site Number : 8400025, Fort Collins, Colorado
  - South Florida Neurology Associates Site Number : 8400029, Boca Raton, Florida
  - MS & Neuromuscular Center of Excellence Site Number : 8400172, Clearwater, Florida
  - University of Florida, Fixel Center for Neurology Site Number : 8400159, Gainesville, Florida
  - Neurology Associates, PA- Site Number : 8400004, Maitland, Florida
  - University of South Florida Site Number : 8400006, Tampa, Florida
  - Velocity Clinical Research Site Number : 8400003, Savannah, Georgia
  - Hawaii Pacific Neuroscience Site Number : 8400103, Honolulu, Hawaii
  - Consultants In Neurology- Site Number : 8400011, Northbrook, Illinois
  - Methodist Hospital Site Number : 8400164, Merrillville, Indiana
  - College Park Family Care Center Site Number : 8400044, Overland Park, Kansas
  - University of Kentucky Site Number : 8400106, Lexington, Kentucky
  - Ochsner Baptist Clinical Trials Unit (CTU)- Site Number : 8400107, New Orleans, Louisiana
  - International Neurorehabilitation Institute Site Number : 8400034, Lutherville, Maryland
  - Tufts Medical Center Site Number : 8400072, Boston, Massachusetts
  - University of Massachusetts Site Number : 8400014, Worcester, Massachusetts
  - Michigan Institute For Neurological Disorders Site Number : 8400058, Farmington Hills, Michigan
  - The Memorial Hospital- Site Number : 8400033, Owosso, Michigan
  - Mayo Clinic Site Number : 8400111, Rochester, Minnesota
  - Sharlin Health & Neurology Site Number : 8400093, Ozark, Missouri
  - University Of Nebraska- Site Number : 8400129, Omaha, Nebraska
  - Hackensack University Hospital Site Number : 8400047, Hackensack, New Jersey
  - University of New Mexico Site Number : 8400032, Albuquerque, New Mexico
  - Icahn School of Medicine at Mount Sinai (Department of Endoc Site Number : 8400038, New York, New York
  - Neurology Associates of Stony Brook Site Number : 8400042, Stony Brook, New York
  - Duke Neurological Disorders Clinic- Site Number : 8400098, Durham, North Carolina
  - Meridian Clinical Research, LLC- Site Number : 8400005, Raleigh, North Carolina
  - Atrium Health Wake Forest Baptist Site Number : 8400116, Winston-Salem, North Carolina
  - Riverhills Neuroscience - Norwood Site Number : 8400167, Cincinnati, Ohio
  - Cleveland Clinic Site Number : 8400125, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center- Site Number : 8400150, Columbus, Ohio
  - The Boster Center for Multiple Sclerosis Site Number : 8400147, Columbus, Ohio
  - Providence Multiple Sclerosis Center Site Number : 8400020, Portland, Oregon
  - Jefferson Neurology Associates Site Number : 8400016, Philadelphia, Pennsylvania
  - Mountain View Clinical Research Site Number : 8400024, Greer, South Carolina
  - Mt Olympus Medical Research Site Number : 8400163, Katy, Texas
  - Neurology Center of San Antonio Site Number : 8400036, San Antonio, Texas
- Argentina (2):
  - Investigational Site Number : 0320002, CABA, Buenos Aires
  - Investigational Site Number : 0320003, Rosario, Santa Fe Province
- Australia (3):
  - Investigational Site Number : 0360005, Concord, New South Wales
  - Investigational Site Number : 0360006, St Leonards, New South Wales
  - Investigational Site Number : 0360003, Hobart, Tasmania
- Austria (2):
  - Investigational Site Number : 0400004, Linz
  - Investigational Site Number : 0400002, Vienna
- Belarus (2):
  - Investigational Site Number : 1120004, Vitebsk
  - Investigational Site Number : 1120005, Vitebsk
- Belgium (5):
  - Investigational Site Number : 0560009, Brussels
  - Investigational Site Number : 0560004, Ghent
  - Investigational Site Number : 0560008, Liège
  - Investigational Site Number : 0560001, Overpelt
  - Investigational Site Number : 0560007, Woluwe-Saint-Lambert
- Brazil (2):
  - Instituto de Neurologia de Curitiba Site Number : 0760002, Curitiba, Paraná
  - CPQuali Pesquisa Clinica Site Number : 0760007, São Paulo, São Paulo
- Bulgaria (5):
  - Investigational Site Number : 1000002, Pleven
  - Investigational Site Number : 1000004, Sofia
  - Investigational Site Number : 1000008, Sofia
  - Investigational Site Number : 1000001, Sofia
  - Investigational Site Number : 1000011, Sofia
- Canada (10):
  - Investigational Site Number : 1240002, Edmonton, Alberta
  - Investigational Site Number : 1240016, Vancouver, British Columbia
  - Investigational Site Number : 1240012, Hamilton, Ontario
  - Investigational Site Number : 1240003, Ottawa, Ontario
  - Investigational Site Number : 1240013, Toronto, Ontario
  - Investigational Site Number : 1240004, Montreal, Quebec
  - Investigational Site Number : 1240015, Montreal, Quebec
  - Investigational Site Number : 1240007, Sherbrooke, Quebec
  - Investigational Site Number : 1240001, Québec
  - Investigational Site Number : 1240021, Québec
- Chile (2):
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
- China (13):
  - Investigational Site Number : 1560003, Beijing
  - Investigational Site Number : 1560012, Beijing
  - Investigational Site Number : 1560009, Beijing
  - Investigational Site Number : 1560025, Beijing
  - Investigational Site Number : 1560004, Changchun
  - Investigational Site Number : 1560015, Changsha
  - Investigational Site Number : 1560005, Chengdu
  - Investigational Site Number : 1560035, Fuzhou
  - Investigational Site Number : 1560002, Guangzhou
  - Investigational Site Number : 1560027, Hohhot
  - Investigational Site Number : 1560001, Shanghai
  - Investigational Site Number : 1560008, Taiyuan
  - Investigational Site Number : 1560026, Wenzhou
- Colombia (2):
  - Investigational Site Number : 1700003, Bogotá
  - Investigational Site Number : 1700001, Bogotá
- Croatia (2):
  - Investigational Site Number : 1910001, Zagreb
  - Investigational Site Number : 1910002, Zagreb
- Czechia (4):
  - Investigational Site Number : 2030002, Brno
  - Investigational Site Number : 2030004, Hradec Králové
  - Investigational Site Number : 2030001, Jihlava
  - Investigational Site Number : 2030003, Teplice
- Denmark (2):
  - Investigational Site Number : 2080001, Esbjerg
  - Investigational Site Number : 2080005, Holstebro
- Investigational Site Number : 2330001, Tallinn, Estonia
- France (13):
  - Investigational Site Number : 2500011, Bron
  - Investigational Site Number : 2500005, Clermont-Ferrand
  - Investigational Site Number : 2500015, Gonesse
  - Investigational Site Number : 2500009, Lille
  - Investigational Site Number : 2500006, Montpellier
  - Investigational Site Number : 2500008, Nancy
  - Investigational Site Number : 2500017, Nîmes
  - Investigational Site Number : 2500014, Paris
  - Investigational Site Number : 2500007, Paris
  - Investigational Site Number : 2500004, Poissy
  - Investigational Site Number : 2500003, Rennes
  - Investigational Site Number : 2500001, Strasbourg
  - Investigational Site Number : 2500012, Toulouse
- Georgia (4):
  - Investigational Site Number : 2680005, Tbilisi
  - Investigational Site Number : 2680009, Tbilisi
  - Investigational Site Number : 2680003, Tbilisi
  - Investigational Site Number : 2680004, Tbilisi
- Germany (13):
  - Investigational Site Number : 2760005, Bayreuth
  - Investigational Site Number : 2760009, Berlin
  - Investigational Site Number : 2760015, Berlin
  - Investigational Site Number : 2760020, Bochum
  - Investigational Site Number : 2760001, Dresden
  - Investigational Site Number : 2760021, Düsseldorf
  - Investigational Site Number : 2760012, Essen
  - Investigational Site Number : 2760002, Giessen
  - Investigational Site Number : 2760006, Hanover
  - Investigational Site Number : 2760018, München
  - Investigational Site Number : 2760008, Münster
  - Investigational Site Number : 2760004, Rostock
  - Investigational Site Number : 2760011, Ulm
- Greece (7):
  - Investigational Site Number : 3000001, Athens
  - Investigational Site Number : 3000006, Athens
  - Investigational Site Number : 3000002, Athens
  - Investigational Site Number : 3000004, Larissa
  - Investigational Site Number : 3000007, Marousi
  - Investigational Site Number : 3000003, Thessaloniki
  - Investigational Site Number : 3000009, Thessaloniki
- Hungary (3):
  - Investigational Site Number : 3480206, Budapest
  - Investigational Site Number : 3480202, Budapest
  - Investigational Site Number : 3480203, Budapest
- India (3):
  - Investigational Site Number : 3560014, Bengaluru
  - Investigational Site Number : 3560004, Mangaluru
  - Investigational Site Number : 3560005, New Delhi
- Israel (3):
  - Investigational Site Number : 3760008, Jerusalem
  - Investigational Site Number : 3760001, Ramat Gan
  - Investigational Site Number : 3760004, Safed
- Italy (9):
  - Investigational Site Number : 3800002, Pozzilli, Isernia
  - Investigational Site Number : 3800007, Cagliari
  - Investigational Site Number : 3800015, Catania
  - Investigational Site Number : 3800018, Chieti
  - Investigational Site Number : 3800016, Florence
  - Investigational Site Number : 3800001, Milan
  - Investigational Site Number : 3800003, Napoli
  - Investigational Site Number : 3800006, Napoli
  - Investigational Site Number : 3800013, Roma
- Japan (15):
  - Investigational Site Number : 3920016, Chiba, Chiba
  - Investigational Site Number : 3920008, Koriyama-shi, Fukushima
  - Investigational Site Number : 3920022, Morioka, Iwate
  - Investigational Site Number : 3920023, Sagamihara-shi, Kanagawa
  - Investigational Site Number : 3920011, Kyoto, Kyoto
  - Investigational Site Number : 3920020, Sendai, Miyagi
  - Investigational Site Number : 3920005, Niigata, Niigata
  - Investigational Site Number : 3920004, Moriguchi-shi, Osaka
  - Investigational Site Number : 3920001, Osaka, Osaka
  - Investigational Site Number : 3920018, Kawagoe-shi, Saitama
  - Investigational Site Number : 3920014, Bunkyo-ku, Tokyo
  - Investigational Site Number : 3920003, Kodaira-shi, Tokyo
  - Investigational Site Number : 3920010, Ōta-ku, Tokyo
  - Investigational Site Number : 3920017, Shinjuku-ku, Tokyo
  - Investigational Site Number : 3920015, Toyama, Toyama
- Investigational Site Number : 4280002, Riga, Latvia
- Mexico (5):
  - Investigational Site Number : 4840004, Guadalajara, Jalisco
  - Investigational Site Number : 4840001, Mexico City, Mexico City
  - Investigational Site Number : 4840005, Mexico City
  - Investigational Site Number : 4840007, Tlalnepantla
  - Investigational Site Number : 4840003, Veracruz
- Netherlands (3):
  - Investigational Site Number : 5280003, Breda
  - Investigational Site Number : 5280006, Groningen
  - Investigational Site Number : 5280002, Sittard-Geleen
- Norway (2):
  - Investigational Site Number : 5780003, Bergen
  - Investigational Site Number : 5780005, Tromsø
- Investigational Site Number : 6040004, Lima, Peru
- Poland (6):
  - Investigational Site Number : 6160003, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Investigational Site Number : 6160001, Lodz, Lódzkie
  - Investigational Site Number : 6160005, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160006, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160007, Katowice, Silesian Voivodeship
  - Investigational Site Number : 6160004, Katowice, Silesian Voivodeship
- Portugal (6):
  - Investigational Site Number : 6200001, Braga
  - Investigational Site Number : 6200007, Lisbon
  - Investigational Site Number : 6200012, Lisbon
  - Investigational Site Number : 6200002, Matosinhos Municipality
  - Investigational Site Number : 6200010, Porto
  - Investigational Site Number : 6200004, Santa Maria da Feira
- Romania (6):
  - Investigational Site Number : 6420008, Bucharest
  - Investigational Site Number : 6420004, Campulung Muscel
  - Investigational Site Number : 6420003, Constanța
  - Investigational Site Number : 6420013, Oradea
  - Investigational Site Number : 6420001, Târgu Mureş
  - Investigational Site Number : 6420002, Timișoara
- Russia (15):
  - Investigational Site Number : 6430018, Barnaul
  - Investigational Site Number : 6430023, Kaliningrad
  - Investigational Site Number : 6430004, Kazan'
  - Investigational Site Number : 6430021, Krasnoyarsk
  - Investigational Site Number : 6430013, Moscow
  - Investigational Site Number : 6430011, Moscow
  - Investigational Site Number : 6430014, Nizhny Novgorod
  - Investigational Site Number : 6430008, Pyatigorsk
  - Investigational Site Number : 6430015, Rostov-on-Don
  - Investigational Site Number : 6430017, Saint Petersburg
  - Investigational Site Number : 6430009, Samara
  - Investigational Site Number : 6430020, Saransk
  - Investigational Site Number : 6430007, Tyumen
  - Investigational Site Number : 6430006, Ufa
  - Investigational Site Number : 6430022, Yekaterinburg
- Serbia (2):
  - Investigational Site Number : 6880001, Belgrade
  - Investigational Site Number : 6880002, Kragujevac
- Investigational Site Number : 7100001, Pretoria, South Africa
- Spain (15):
  - Investigational Site Number : 7240012, A Coruña, A Coruña [La Coruña]
  - Investigational Site Number : 7240015, Santiago de Compostela, A Coruña [La Coruña]
  - Investigational Site Number : 7240007, Seville, Andalusia
  - Investigational Site Number : 7240010, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240013, Bilbao, Bizkaia
  - Investigational Site Number : 7240011, Salt, Girona [Gerona]
  - Investigational Site Number : 7240016, Las Palmas de Gran Canaria, Las Palmas
  - Investigational Site Number : 7240002, Majadahonda, Madrid
  - Investigational Site Number : 7240001, Pozuelo de Alarcón, Madrid
  - Investigational Site Number : 7240004, Córdoba
  - Investigational Site Number : 7240003, Madrid
  - Investigational Site Number : 7240005, Málaga
  - Investigational Site Number : 7240006, Murcia
  - Investigational Site Number : 7240014, Palma de Mallorca
  - Investigational Site Number : 7240008, Valencia
- Sweden (2):
  - Investigational Site Number : 7520001, Gothenburg
  - Investigational Site Number : 7520005, Motala
- Investigational Site Number : 7640001, Bangkok, Thailand
- Turkey (Türkiye) (15):
  - Investigational Site Number : 7920009, Ankara
  - Investigational Site Number : 7920014, Ankara
  - Investigational Site Number : 7920005, Eskişehir
  - Investigational Site Number : 7920010, Hatay
  - Investigational Site Number : 7920016, Istanbul
  - Investigational Site Number : 7920003, Istanbul
  - Investigational Site Number : 7920002, Istanbul
  - Investigational Site Number : 7920007, Istanbul
  - Investigational Site Number : 7920015, Izmir
  - Investigational Site Number : 7920018, Izmir
  - Investigational Site Number : 7920001, İzmit
  - Investigational Site Number : 7920017, Konya
  - Investigational Site Number : 7920011, Kütahya
  - Investigational Site Number : 7920012, Mersin
  - Investigational Site Number : 7920013, Samsun
- Ukraine (13):
  - Investigational Site Number : 8040020, Chernivtsi
  - Investigational Site Number : 8040012, Ivano-Frankivsk
  - Investigational Site Number : 8040017, Kharkiv
  - Investigational Site Number : 8040025, Kharkiv
  - Investigational Site Number : 8040023, Kharkiv
  - Investigational Site Number : 8040014, Kyiv
  - Investigational Site Number : 8040013, Kyiv
  - Investigational Site Number : 8040015, Kyiv
  - Investigational Site Number : 8040011, Lutsk
  - Investigational Site Number : 8040002, Lviv
  - Investigational Site Number : 8040007, Lviv
  - Investigational Site Number : 8040010, Odesa
  - Investigational Site Number : 8040024, Vinnytsia
- United Kingdom (11):
  - Investigational Site Number : 8260003, Exeter, Devon
  - Investigational Site Number : 8260016, Canterbury, Kent
  - Investigational Site Number : 8260006, London, London, City of
  - Investigational Site Number : 8260005, London, London, City of
  - Investigational Site Number : 8260010, Swansea, Neath Port Talbot
  - Investigational Site Number : 8260012, Nottingham, Nottinghamshire
  - Investigational Site Number : 8260013, Oxford, Oxfordshire
  - Investigational Site Number : 8260001, Cardiff, Vale of Glamorgan, the
  - Investigational Site Number : 8260009, Bristol
  - Investigational Site Number : 8260019, Salford
  - Investigational Site Number : 8260007, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC16035 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25239&tenant=MT_SNY_9011